CLINICAL TRIAL: NCT01841528
Title: Live Birth After Fresh Embryo Transfer vs Elective Embryo Cryopreservation/Frozen Embryo Transfer in Women With Polycystic Ovary Syndrome Undergoing IVF: A Multi-center Prospective Randomized Clinical Trial
Brief Title: Live Birth After Fresh Embryo Transfer Vs Frozen-thawed Embryo Transfer in Women With Polycystic Ovary Syndrome
Acronym: FreFro-PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zi-jiang Chen (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Anhui Medical University (Other); RenJi Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); LanZhou University (Other); Guangxi provincial maternal and chidren's hospital (Unknown); Renmin Hospital of Wuhan University (Other); Yantai Yuhuangding Hospital (Other); Jiangxi Maternal and Child Health Hospital (Other); Sir Run Run Shaw Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Reproductive Medicine Center in Shenyang City (Unknown)
Responsible Party: Sponsor-Investigator, Zi-jiang Chen, Director of Reproductive medical center of Shandong University, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDUIVF001
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: Polycystic Ovary Syndrome; Infertility; In-vitro fertilization; fresh embryo transfer; frozen-thawed embryo transfer
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fresh embryo transfer group (Experimental): rFSH/GnRH antagonist will be administered for ovarian stimulation. Two fresh embryos will be transferred at Day 3. Luteal phase support will last 2 weeks for all subjects in this group. Two weeks after embryo transfer, serum human chorionic gonadotropin (HCG) will be measured to determine pregnant or not. If biochemical pregnancy is achieved, luteal phase support will be continued to 10 weeks gestation. Pregnancy complications and final outcome will be followed up till 6 weeks after delivery.
  Interventions: Other: fresh embryo transfer
- frozen-thawed embryo transfer group (Experimental): rFSH/GnRH antagonist will be administered for ovarian stimulation. All embryos will be vitrified in fresh cycle, and at least 2 embryos should be frozen at Day 3. Two months later, two thawed Day 3 embryos will be transferred with hormone replacement therapy (HRT) prepared endometrium. Luteal phase support will last 2 weeks for all subjects in this group. Two weeks after embryo transfer, serum human chorionic gonadotropin (HCG) will be measured to determine pregnant or not. If biochemical pregnancy is achieved, luteal phase support will be continued to 10 weeks gestation. Pregnancy complications and final outcome will be followed up till 6 weeks after delivery.
  Interventions: Other: frozen-thawed embryo transfer

INTERVENTIONS:
Other: fresh embryo transfer — rFSH/GnRH antagonist will be administered for ovarian stimulation. Oocyte pick-up will be performed when at least two follicles ≥18mm. Two fresh embryos will be transferred at Day 3. Luteal phase support will last 2 weeks for all subjects in this group. Two weeks after embryo transfer, serum HCG will be measured to determine pregnant or not. If biochemical pregnancy is achieved, luteal phase support will be continued to 10 weeks gestation. Pregnancy complications and final outcome will be followed up till 6 weeks after delivery.
  Arms: fresh embryo transfer group
Other: frozen-thawed embryo transfer — rFSH/GnRH antagonist will be administered for ovarian stimulation. Oocyte pick-up will be performed when at least two follicles ≥18mm. All embryos will be vitrified in fresh cycle, and at least 2 embryos should be frozen at Day 3. Two months later, two thawed Day 3 embryos will be transferred with HRT (hormone replacement therapy) prepared endometrium. Luteal phase support will last 2 weeks for all subjects in this group. Two weeks after embryo transfer, serum HCG will be measured to determine pregnant or not. If biochemical pregnancy is achieved, luteal phase support will be continued to 10 weeks gestation. Pregnancy complications and final outcome will be followed up till 6 weeks after delivery.
  Arms: frozen-thawed embryo transfer group

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine disorders in women of childbearing age. However, the optimal infertility treatment for PCOS patients is still a matter of controversy. Despite producing more follicles and more oocytes than other women undergoing controlled ovarian hyperstimulation during an IVF cycle, women with PCOS have comparable or lower pregnancy rates. Additionally women with PCOS patients undergoing IVF have a higher risk of developing ovarian hyperstimulation syndrome (OHSS), which may be aggravated by pregnancy after an embryo transfer in a fresh cycle. Further women with PCOS are thought to have higher rates of later pregnancy complications including spontaneous abortion, pre-eclampsia, and preterm labor that may be related to impaired implantation in the superovulated endometrium. We propose a randomized clinical trial of elective embryo cryopreservation followed by a programmed cycle of endometrial preparation and frozen embryo transfer (FET) compared to fresh embryo transfer in women with PCOS undergoing in vitro fertilization (IVF).

DETAILED DESCRIPTION:
This will be a multi-center, prospective, randomized (1:1 ratio)clinical trial of frozen-thawed embryo transfer vs. fresh embryo transfer after a uniform gonadotropin-releasing hormone (GnRH) antagonist protocol in infertile PCOS patients receiving IVF therapy. Qualified 1180 patients are randomized into either of two groups: group A will undergo fresh embryo transfer (590 cases), Group B will undergo elective cryopreservation of all embryos followed by transfer of thawed embryos to a programmed endometrium (590 cases). All of the participants will receive recombinant follicule stimulating hormone (rFSH)/GnRH antagonist protocol for ovarian stimulation and standardized luteal phase support.

The target population will be infertile PCOS patients aged between 20 and 35 years, diagnosed by the Chinese PCOS Criteria(i.e. menstrual disorders PLUS either one of the remaining two criteria, hyperandrogenism or polycystic ovaries on ultrasound, with exclusion of secondary causes of hyperandrogenism and ovulation dysfunction). And subjects will be those who are undergoing their first IVF or intracytoplasmatic sperm injection (ICSI) cycle without other known factors interfere reproductive or metabolic functions.

The randomization will take place at the oocyte pick-up day by an on-line randomization system.

The pregnancy test results, pregnancy complications, congenital anomalies neonatal complications will be followed up by checking medical records and telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed as PCOS according to Chinese PCOS diagnosis criteria;
* Women who have ≥1 years history of infertility;
* Women aged ≥20 and <35 years old;
* Women with body weight ≥40kg;
* Women who have at least one of the following indications for IVF or ICSI:

  1. Ovulation dysfunction and failed to become pregnant from ovulation induction treatment;
  2. Tubal factors: unilateral or bilateral tubal obstruction, adhesion, unilateral or bilateral Salpingectomy or tubal ligation;
  3. Male factors: oligoasthenozoospermia, obstructive azoospermia;
* Women who are undergoing their first cycle of IVF or ICSI;
* Women who retrieved oocytes number > 3;
* Women who are capable of giving informed consent.

Exclusion Criteria:

* Women who underwent unilateral ovariectomy;
* Women diagnosed as uterus abnormality: malformed uterus (uterus unicorns, septate uterus, duplex uterus, uterus bicomis), adenomyosis, submucous myoma, intrauterine adhesion;
* Women or their partner with abnormal chromosome karyotype including chromosome polymorphism;
* Women who have experienced recurrent spontaneous abortion (including biochemical pregnancy abortion) more than 2 times;
* Women with medical condition that represent contraindication to assisted reproductive technology and/or pregnancy;
* Women who has developed severe OHSS before oocyte pick-up day;
* Women with retrieved oocytes number ≤3;
* Women who are unable to comply with the study procedures.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1180 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 10 months for group A, 12 months for group B
  This will be based on the outcome of either the fresh embryo transfer after ovarian stimulation (Group A) or the outcome of the first frozen embryo transfer cycle (Group B) as will all other secondary outcomes.

SECONDARY OUTCOMES:
Ovarian hyperstimulation syndrome (OHSS) incidence | 2 months in maximum estimated
clinical pregnancy rate | 35 days after embryo transfer
  This will be based on the visualization of a intrauterine gestational sac by ultrasound.
Pregnancy Loss rate | 28 weeks gestation in maximum
  Loss of pregnancy will be defined by any positive pregnancy test that does not result in a live birth and will be tracked.
ectopic pregnancy rate | 7~8 weeks gestation
singleton live birth rate | 10 months for group A, 12 months for group B
pregnancy complication rate | 10 months for group A, 12 months for group B
  Complications of pregnancy including gestational hypertension, diabetes, preterm labor, disorders of placentation will be collected in all patients with ongoing clinical pregnancies.
Congenital Anomalies rate | 10 months for group A, 12 months for group B
  We will collect all recognized fetal and infant anomalies that occur within the trial.
neonatal complication rate | within one month after labor
  We will collect complications that occur in the neonate including admission to the neonatal intensive care unit (NICU), hospitalization, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zi-jiang Chen, MD, Principal Investigator — Repreductive medical hospital affiliated to Shandong University
Locations (14):
- China (14):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangxi Maternal and Child Health Hospital, Nanning, Guangxi
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Reproductive Medicine Center in Shenyang City, Shenyang, Liaoning
  - Reproductive medical hospital affiliated to Shandong University, Jinan, Shandong
  - Yuhuangding Hospital in Yantai, Yantai, Shandong
  - Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial Maternity and Children's Hospital, Xi’an, Shanxi
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] [1] Boomsma CM, Eijkemans MJ, Hughes EG, et al. A meta-analysis of pregnancy outcomes in women with polycystic ovary syndrome. Hum Reprod Update 12:673-83,2006. [2] Hayashi M, Nakai A, Satoh S, et al. Adverse obstetric and perinatal outcomes of singleton pregnancies may be related to maternal factors associated with infertility rather than the type of assisted reproductive technology procedure used. Fertil Steril 98:922-928,2012. [3] Chen XK, Wen SW, Bottomley J, et al. In vitro fertilization is associated with an increased risk for preeclampsia. Hypertens Pregnancy 28:1-12,2009. [4] Thomopoulos C, Tsioufis C, Michalopoulou H, et al. Assisted reproductive technology and pregnancy-related hypertensive complications: a systematic review. J Hum Hypertens 27:148-57,2013. [5] Haavaldsen C, Tanbo T, Eskild A. Placental weight in singleton pregnancies with and without assisted reproductive technology: a population study of 536,567 pregnancies. Hum Reprod 27:576-82,2012. [6] Maheshwari A, Pandey S, Shetty A, et al. Obstetric and perinatal outcomes in singleton pregnancies resulting from the transfer of frozen thawed versus fresh embryos generated through in vitro fertilization treatment: a systematic review and meta-analysis. Fertil Steril 98:368-77 e1-9,2012. [7] Kalra SK, Ratcliffe SJ, Coutifaris C, et al. Ovarian stimulation and low birth weight in newborns conceived through in vitro fertilization. Obstet Gynecol 118:863-871,2011.
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543
- [Derived] Wei D, Yu Y, Sun M, Shi Y, Sun Y, Deng X, Li J, Wang Z, Zhao S, Zhang H, Legro RS, Chen ZJ. The Effect of Supraphysiological Estradiol on Pregnancy Outcomes Differs Between Women With PCOS and Ovulatory Women. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2735-2742. doi: 10.1210/jc.2018-00613. PMID 29718297
- [Derived] Zhang B, Wei D, Legro RS, Shi Y, Li J, Zhang L, Hong Y, Sun G, Zhang T, Li W, Chen ZJ. Obstetric complications after frozen versus fresh embryo transfer in women with polycystic ovary syndrome: results from a randomized trial. Fertil Steril. 2018 Feb;109(2):324-329. doi: 10.1016/j.fertnstert.2017.10.020. Epub 2018 Jan 17. PMID 29338857
- [Derived] Wei D, Zhang B, Shi Y, Zhang L, Zhao S, Du Y, Xu L, Legro RS, Zhang H, Chen ZJ. Effect of Preconception Impaired Glucose Tolerance on Pregnancy Outcomes in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3822-3829. doi: 10.1210/jc.2017-01294. PMID 28938429
- [Derived] Wei D, Shi Y, Li J, Wang Z, Zhang L, Sun Y, Zhou H, Xu Y, Wu C, Liu L, Wu Q, Zhuang L, Du Y, Li W, Zhang H, Legro RS, Chen ZJ. Effect of pretreatment with oral contraceptives and progestins on IVF outcomes in women with polycystic ovary syndrome. Hum Reprod. 2017 Feb;32(2):354-361. doi: 10.1093/humrep/dew325. Epub 2016 Dec 19. PMID 27999118
- [Derived] Chen ZJ, Shi Y, Sun Y, Zhang B, Liang X, Cao Y, Yang J, Liu J, Wei D, Weng N, Tian L, Hao C, Yang D, Zhou F, Shi J, Xu Y, Li J, Yan J, Qin Y, Zhao H, Zhang H, Legro RS. Fresh versus Frozen Embryos for Infertility in the Polycystic Ovary Syndrome. N Engl J Med. 2016 Aug 11;375(6):523-33. doi: 10.1056/NEJMoa1513873. PMID 27509101
- [Derived] Shi Y, Wei D, Liang X, Sun Y, Liu J, Cao Y, Zhang B, Legro RS, Zhang H, Chen ZJ. Live birth after fresh embryo transfer vs elective embryo cryopreservation/frozen embryo transfer in women with polycystic ovary syndrome undergoing IVF (FreFro-PCOS): study protocol for a multicenter, prospective, randomized controlled clinical trial. Trials. 2014 May 2;15:154. doi: 10.1186/1745-6215-15-154. PMID 24885793